CLINICAL TRIAL: NCT02593123
Title: Adoptive Immunotherapy in Patients With Relapsed Hematological Malignancy: Effect of Duration and Intensity of Early GVHD Prophylaxis on Long-Term Clinical Outcomes
Brief Title: Adoptive Immunotherapy in Relapsed Hematological Malignancy: Early GVHD Prophylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Massey Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14-10739; HM20005586 (Other: VCU Office of Research Subjects Protection)
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Hodgkin's Lymphoma; Lymphoid Leukemia; Lymphoma; Leukemia; Myeloma; Acute Lymphocytic Leukemia; Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Multiple Myeloma; Chronic Myelogenous Leukemia; Myelodysplastic Syndromes; Recurrent Acute Myeloid Leukemia, Adult; Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia
Keywords: Donor Type (Matched Related Donor or Matched Unrelated Donor)
MeSH Terms: conditions — Hodgkin Disease; Leukemia, Lymphoid; Lymphoma; Leukemia; Neoplasms, Plasma Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Mycophenolic Acid; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (MMF-15, sargramostim) (Experimental): Patients receive mycophenolate mofetil (MMF) PO or IV twice daily (BID) on days 0-15 and sargramostim SC from post-transplant day 4 until neutrophil engraftment.
  Interventions: Drug: mycophenolate mofetil; Biological: Sargramostim
- Arm II (MMF-30, filgrastim) (Active Comparator): Patients receive mycophenolate mofetil PO or IV (twice daily) BID on days 0-30 and filgrastim G-CSF from post-transplant day 4 until neutrophil engraftment.
  Interventions: Drug: mycophenolate mofetil; Biological: Filgrastim

INTERVENTIONS:
Drug: mycophenolate mofetil — Given PO, by mouth, orally or IV, intravenous medication administration.
  Other Names: CellCept
Biological: Sargramostim — GM-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-15 cohort will receive sargramostim (GM-CSF) 250 mcg/m2/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
  Patients receiving GM-CSF will also receive inhaled corticosteroids, fluticasone (Flovent) 2 puffs twice daily, starting on post-transplant day 4 and stopping after cessation of GM-CSF, to diminish the risk of pneumonitis.
  Note: At investigator discretion, patients in the MMF-15 cohort who have preexisting pulmonary risk factors, will be permitted to receive G-CSF.
  Other Names: GM-CSF; colony stimulating factor 2; CSF2; granulocyte macrophage colony stimulating factor
  Arms: Arm I (MMF-15, sargramostim)
Biological: Filgrastim — G-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-30 cohort will receive filgrastim (G-CSF) 5 mcg/kg/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
  Other Names: G-CSF; GCSF; colony-stimulating factor 3; CSF 3; granulocyte colony stimulating factor
  Arms: Arm II (MMF-30, filgrastim)

SUMMARY:
Determine the relapse-free, donor lymphocyte infusion (DLI)-free survival in patients receiving the investigational regimen.This is a randomized phase II clinical trial, comparing two different dosing schedules of mycophenolate mofetil for graft versus host disease (GVHD) prevention following allogeneic stem cell transplantation. Risk for relapse, GVHD and non-relapse mortality will be assessed. Adaptive randomization between two study arms will be performed based on T cell counts at day 60.

DETAILED DESCRIPTION:
In this study, the investigators will utilize a regimen combining low dose total body irradiation and rabbit ATG to facilitate stem cell transplantation (SCT) with human leukocyte antigen (HLA) matched related and unrelated donors. Based on the hypothesis that early treatment interventions have significant late effects in allogeneic SCT, a simple intervention, varying the duration of intense immunosuppression following SCT, will be investigated in this study. This may allow more robust recovery of donor immune system cells in the first two months following transplantation and eventually result in lower risk of cancer relapse, while maintaining effective graft versus host disease (GVHD) control. Patients will be randomly assigned to receive GVHD prevention therapy using one of two different immunosuppressive regimens with tacrolimus & mycophenolate mofetil (MMF). Patients assigned to the investigational group will receive MMF for 15 days following SCT with growth factor support using granulocyte macrophage colony stimulating factor (GM-CSF) beginning on post-transplant day 4. Patients randomized to the standard treatment group will receive MMF for 30 days following SCT with cytokine support using granulocyte colony stimulating factor (G-CSF) beginning on post-transplant day 4. If one of these treatment groups demonstrates an improvement in donor immune cell recovery, there may be a slow increase in the likelihood of patients being assigned to that more successful treatment group. Eventually the two groups will be compared with respect to the likelihood of either relapse or GVHD developing.

ELIGIBILITY:
Inclusion Criteria

* Any of the following high risk or recurrent hematological malignancies:
* Hodgkin lymphoma (HL)
* Non-Hodgkin lymphoma (NHL)
* Chronic lymphocytic leukemia (CLL)
* Multiple myeloma (MM)
* Acute myelogenous leukemia (AML)
* Acute lymphocytic leukemia (ALL)
* Chronic myelogenous leukemia (CML)
* Myelodysplastic syndrome (MDS)

  *Note: Determination that the malignancy is high risk will be made by the investigator.
* Investigator determination that the patient is an appropriate candidate for reduced intensity allogeneic SCT with the standard Massey Cancer Center-Virginia Commonwealth Health System Bone Marrow Transplant Massey Cancer Center Virginia Commonwealth University Health System Bone Marrow Transplant (MCC-VCUHS BMT) Program regimen employed in this trial
* Patients with or without previous myeloablative autologous transplant
* HLA-matched stem cell donor, either related (6/6 or 5/6 loci matched) or unrelated (8/8 or 7/8 loci matched)

  *Note: Unrelated donors must be matched at HLA-A, -B, -C, and -DRB1 loci. However, a single locus mismatch will be acceptable in the event a more closely matched donor is not available.
* Age ≥ 40 to < 75 years; patients 18 to 39 years of age will be eligible only if the investigator has determined that the patient has comorbidity(ies) precluding conventional allogeneic transplantation with full intensity myeloablative conditioning
* Karnofsky Performance Status of 70-100%
* Negative serology for HIV
* Women who are not postmenopausal or have not undergone hysterectomy must have a documented negative serum pregnancy test per standard MCC-VCUHS BMT Program guidelines
* Ability to understand and the willingness to sign a written informed consent document *Note: The consent form must be signed and dated prior to initiation of SCT preparative treatments.

Exclusion Criteria

* Previous therapeutic radiation therapy (RT) that exceeds critical structure tolerance doses as determined by a radiation oncologist
* Uncontrolled viral, fungal, or bacterial infection
* Active meningeal or central nervous system disease
* Previous therapy with rabbit anti-thymocyte globulin (ATG); previous treatment with equine ATG is allowed if more than 3 months ago

  *Note: Previous myeloablative autologous transplant is permitted but not required.
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Toor, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (MMF-15, Sargramostim): Patients receive mycophenolate mofetil (MMF) PO or IV BID on days 0-15 and sargramostim SC from post-transplant day 4 until neutrophil engraftment.
  mycophenolate mofetil: Given PO, by mouth, orally or IV, intravenous medication administration.
  Sargramostim: GM-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-15 cohort will receive sargramostim (GM-CSF) 250 mcg/m2/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
  Patients receiving GM-CSF will also receive inhaled corticosteroids, fluticasone (Flovent) 2 puffs twice daily, starting on post-transplant day 4 and stopping after cessation of GM-CSF, to diminish the risk of pneumonitis.
  Note: At investigator discretion, patients in the MMF-15 cohort who have preexisting pulmonary risk factors, will be permitted to receive G-CSF.
- Arm II (MMF-30, Filgrastim): Patients receive mycophenolate mofetil PO or IV BID on days 0-30 and filgrastim G-CSF from post-transplant day 4 until neutrophil engraftment.
  mycophenolate mofetil: Given PO, by mouth, orally or IV, intravenous medication administration.
  Filgrastim: G-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-30 cohort will receive filgrastim (G-CSF) 5 mcg/kg/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
Period: Overall Study
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Started | 18 | 13
Completed | 15 | 11
Not Completed | 3 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Relapse | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm II (MMF-30, Filgrastim): Patients receive mycophenolate mofetil PO or IV BID on days 0-30 and filgrastim GCSF from post-transplant day 4 until neutrophil engraftment.
  mycophenolate mofetil: Given PO, by mouth, orally or IV, intravenous medication administration.
  Filgrastim: G-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-30 cohort will receive filgrastim (G-CSF) 5 mcg/kg/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
- Total: Total of all reporting groups
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim) | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 10 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Relapse-free/Donor Lymphocyte Infusion(DLI)-Free Survival Rates Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort).
Description: The primary outcome in this study is event-free survival, where the conditional events are the occurrence of relapse DLI.
Time Frame: Up to 2 years following stem cell transplant
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (MMF-15, Sargramostim): Patients receive mycophenolate mofetil (MMF) PO or IV twice daily (BID) on days 0-15 and sargramostim subcutaneous (SC) from post-transplant day 4 until neutrophil engraftment.
  mycophenolate mofetil: Given PO, by mouth, orally or IV, intravenous medication administration.
  Sargramostim: GM-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-15 cohort will receive sargramostim (GM-CSF) 250 mcg/m2/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
  Patients receiving GM-CSF will also receive inhaled corticosteroids, fluticasone (Flovent) 2 puffs twice daily, starting on post-transplant day 4 and stopping after cessation of GM-CSF, to diminish the risk of pneumonitis.
  Note: At investigator discretion, patients in the MMF-15 cohort who have preexisting pulmonary risk factors, will be permitted to receive G-CSF.
- Arm II (MMF-30, Filgrastim): Patients receive mycophenolate mofetil PO or IV twice daily (BID) on days 0-30 and filgrastim from post-transplant day 4 until neutrophil engraftment.
  mycophenolate mofetil: Given PO, by mouth, orally or IV, intravenous medication administration.
  Filgrastim: G-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-30 cohort will receive filgrastim (G-CSF) 5 mcg/kg/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
Participants
  Event Free Survival Yes | 7 | 4
  Event Free Survival No | 8 | 7

2. Secondary Outcome: The Difference Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort) Day 60 Donor-derived (dd) Cluster of Differentiation (CD)3 10E3per microL Counts.
Description: Day 60 donor-derived (dd) cluster of differentiation (CD)3 counts measured by 10E3per microL.
Time Frame: 60 Days Following Stem Cell Transplant
Measure: Mean (Standard Error); unit: 10^3 *cells* per microliter
Groups:
- Arm II (MMF-30, Filgrastim): Patients receive mycophenolate mofetil PO or IV BID on days 0-30 and filgrastim from post-transplant day 4 until neutrophil engraftment.
  mycophenolate mofetil: Given PO, by mouth, orally or IV, intravenous medication administration.
  Filgrastim: G-CSF beginning post-transplant day 4 and continuing until hematopoietic reconstitution. Patients in the MMF-30 cohort will receive filgrastim (G-CSF) 5 mcg/kg/day beginning on post-transplant day 4 and continuing until neutrophil engraftment.
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
10^3 *cells* per microliter | 383.0 (539) | 254.1 (375)

3. Secondary Outcome: The Probability of Overall Survival (OS) Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort)
Description: Overall survival (days to event or survival: time-to-event; survival: categorical)
Time Frame: Randomization up to 2 years
Measure: Number; unit: Probablility of 2 year survival
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 9
Probablility of 2 year survival | 0.78 | 0.5

4. Secondary Outcome: Differences Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort) With Acute Graft Vs Host Disease (GVHD)
Description: The number of patients diagnosed with acute acute GVHD between patients randomized to MMF-30 (control cohort) and MMF-15 (investigational cohort)
Time Frame: 60 Days following stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
Participants | 4 | 8

5. Secondary Outcome: Differences Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort) Diagnosed With Chronic Graft vs Host Disease (GVHD)
Description: The differences in the rates of chronic GVHD between patients randomized to MMF-30 (control cohort) and MMF-15 (investigational cohort)
Time Frame: 60 Days following stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
Participants | 9 | 7

6. Secondary Outcome: Differences Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort) Diagnosed With Opportunistic Infections
Description: The number of patients diagnosed with an opportunistic infections.
Time Frame: 60 Days following stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
Participants | 7 | 9

7. Secondary Outcome: Determine the Differences Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort) With Diagnosis of Engraftment Loss.
Description: Number of patients with engraftment loss.
Time Frame: 60 Days Following Stem Cell Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
Participants | 0 | 1

8. Secondary Outcome: Differences Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort)Diagnosed With Differences in the Rates of Engraftment Syndrome.
Description: Number of patients diagnosed with engraftment syndrome.
Time Frame: 60 Days Following Stem Cell Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
Participants | 0 | 0

9. Secondary Outcome: Differences in the Rates of Achieving Donor Chimerisms (the Percentage of DNA in the Sample Which Comes From the Donor) Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort).
Description: Number of patients that achieved donor chimerisms by day 100.
Time Frame: 100 Days following Stem Cell Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
Participants | 15 | 11

10. Secondary Outcome: Differences in the Rates of T-cell Recovery Kinetics Following Stem Cell Transplantation (SCT) Between Patients Randomized to MMF-30 (Control Cohort) and MMF-15 (Investigational Cohort).
Description: Number of T Cells 10E3 per microL per arm indicating rates of T-cell recovery by Day 100 following SCT.
Time Frame: 100 Days Following Stem Cell Transplantation
Measure: Mean (Standard Deviation); unit: 10^3 *cells* per microliter
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
Number analyzed (Participants) | 15 | 11
10^3 *cells* per microliter | 313.6 (56.5) | 222.2 (81.3)

ADVERSE EVENTS:
Time Frame: All Cause Mortality assessed for 2 years. Serious Adverse Events (SAE's) and Adverse Events (AE's) (Other, not included serious) assessed for 6 months.
Arm/Group | Arm I (MMF-15, Sargramostim) | Arm II (MMF-30, Filgrastim)
All-Cause Mortality (participants affected / at risk) | 4/15 | 6/11
Serious Adverse Events (participants affected / at risk) | 15/15 | 11/11
Other Adverse Events (participants affected / at risk) | 15/15 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MMF-15, Sargramostim) (N=15) | Arm II (MMF-30, Filgrastim) (N=11)
Lung Infection (Infections and infestations) | 2 (2) | 1 (1)
Catheter Infection (Infections and infestations) | 3 (3) | 2 (2)
cardiac disorders, other (Cardiac disorders) | 1 (1) | 0 (0)
surgical and medical procedures, other (Surgical and medical procedures) | 1 (1) | 0 (0)
abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Alanine Aminotransferase (Investigations) | 0 (0) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Entercolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Ileal Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Small Intestine Infection (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MMF-15, Sargramostim) (N=15) | Arm II (MMF-30, Filgrastim) (N=11)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (12) | 4 (7)
neutropenia (Blood and lymphatic system disorders) | 7 (9) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (12) | 5 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 5 (6)
CD4 Lymphocytes Decreased (Investigations) | 1 (1) | 2 (2)
White Blood Cell Count Decreased (Infections and infestations) | 1 (1) | 3 (4)
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Catheter Related Infection (Infections and infestations) | 1 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 6 (6) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT02593123/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT02593123/ICF_001.pdf